CLINICAL TRIAL: NCT05542147
Title: Physiopathological Study of Genetic Modulation of Cardiovascular Effect of PPAR-Alpha Activation (MAGNETIC-PPARA)
Brief Title: Genetic-Dependent Cardiovascular Response to PPAR-Alpha Agonist Fenofibrate
Acronym: MAGNETIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Luca Morieri (Other)
Responsible Party: Sponsor-Investigator, Mario Luca Morieri, Principal Investigator, University Hospital Padova
Organization: University Hospital Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AOP2225
Record Dates: First submitted 2022-09-08; First posted 2022-09-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases; Pharmacogenomic Drug Interaction
Keywords: Diabetes; Precision Medicine; Inflammatory Response; arterial stifness; Endothelial Dysfunction; Lipid profile; Pharmacogenomic Drug Interaction; statins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single-blinded for treatment (Participant), double-blinded for genetics (Participant and Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fenofibrate (Experimental): 1 tablet per day per 12 weeks
  Interventions: Drug: Fenofibrate 145 mg
- Placebo (Placebo Comparator): 1 tablet per day per 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate 145 mg — 1 tablet per day
  Other Names: Fenofibrate
  Arms: Fenofibrate
Drug: Placebo — 1 tablet per day
  Arms: Placebo

SUMMARY:
Fenofibrate, a peroxisome proliferator-activated receptor-alpha (PPAR-a) agonist known to improve diabetic dyslipidemia, has been proposed as a drug to prevent cardiovascular disease (CVD) in type 2 diabetes (T2D). However, the results of clinical trials have been mixed. Supporting the hypothesis that these disappointing results hide a genetic heterogeneity in the CVD response to fenofibrate, a common genetic variant (rs6008845) in the gene coding for PPAR-a has been found to dramatically influence the ability of this drug to reduce CVD events in the ACCORD Lipid trial (PMID:31974142).

The aim of this study is to validate these findings by dissecting the pathways and mechanism through which this variant exerts such a modulatory effect, by means of a randomized clinical trial.

If successful, this project will pave the way to a precision medicine approach to prescribe fenofibrate optimally, offering a cardio-protective drug to those patients that are most likely to experience a robust benefit from this medication.

DETAILED DESCRIPTION:
The main hypothesis of this study is that underlying genetic heterogeneity in the CV response to fibrates can successfully identify subjects with a consistent benefit from this treatment. Supporting this postulate a common genetic variant (rs6008845) in the gene coding for PPAR-alpha has been found to dramatically influence the ability of this drug to reduce CVD events.

This genetic modulation of fenofibrate effectiveness has been found in whites, validated in black participants in the ACCORD Lipid trial, and then replicated in external cohorts. Interestingly, the genetic effect was independent of fenofibrate-induced changes in plasma lipids, suggesting a more complex mechanism of action of fibrates. (PMID:31974142).

Through this randomized study, subjects carrying the different rs6008845 genotypes (TT, TC, CC) will be randomized to receive fenofibrate or placebo for 12 weeks.

The specific aims are:

* To replicate the previous "rs6008845 by fenofibrate" interaction on MACE, testing the fenofibrate-induced changes in endothelial function, arterial stiffness, and markers of endothelium damage.
* To evaluate whether the fenofibrate-induced change on circulating biomarkers is modulated by rs6008845 genotypes. This will provide insight into the mechanism(s) behind the rs6008845 modulation of fenofibrate effectiveness by the identification of circulating biomarkers mirroring this genetic effect. Different known actions of fenofibrate, beyond lipid-lowering effects, such as fenofibrate anti-inflammatory and anti-platelet effects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with previous cardiovascular events or at least one CV risk factor (hypertension, obesity, smoke, age>65 years)
* HbA1c < 8%
* Triglycerides < 200 mg/dl
* On statin treatments and with LDLcholesterol < 100 mg/dl or at maximum statin-tolerated dose
* European ancestry (rational: given the relatively small sample size and the ancestry-differences in allele frequency of rs6008845 T allele [i.e. from 65% in whites to 20% in blacks subjects) this criteria allows to limit ethnic-confounding factors that would reduce the probability of success of this physiopathological study aiming to dissect the mechanism of the genetic modulation of fenofibrate effectiveness).

Exclusion Criteria:

* CKD III stage with eGFR<60 ml/min/1.73
* Uncontrolled hypertension with systolic blood pressure > 170 mmHg at enrollment.
* Hereditary muscle disorders
* Uncontrolled hypothyroidism
* Elevated alcohol consumption
* Hepatic failure
* Allergy to fenofibrate or excipients
* Acute / chronic pancreatitis
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | baseline and 12 weeks
  Differences in fenofibrate induced-changes in Reactive Hyperemia Index (RHI) across rs6008845 genotypes. [RHI is a non-invasive measure of endothelial function, and it is inversely associated with risk of cardiovascular disease].

SECONDARY OUTCOMES:
Arterial Stiffness - Pulse Wave Velocity (PWV) | baseline and 12 weeks
  Differences in fenofibrate induced-changes in PWV across rs6008845 genotypes. [PWV is directly associated with risk of cardiovascular disease]
Endothelial progenitor cells (EPCs) | baseline and 12 weeks
  Differences in fenofibrate induced-changes in circulating levels of EPC across rs6008845 genotypes.
Inflammatory markers and chemokines | baseline and 12 weeks
  Differences in fenofibrate induced-changes in CCL11, CCL27 sVCAM, sE-Selectin, Endothelin-1 across rs6008845 genotypes.
Platelet aggregation induced by adenosine diphosphate (ADP) | baseline and 12 weeks
  Anti-platelet effects will be evaluated as the differences in fenofibrate induced-changes in platelet aggregation induced by adenosine diphosphate (ADP) (i.e. ADPtest) across rs6008845 genotypes.
Platelet aggregation induced by arachidonic acid | baseline and 12 weeks
  Anti-platelet effects will be evaluated as the differences in fenofibrate induced-changes in platelet aggregation induced by arachidonic acid (ASPI test) across rs6008845 genotypes.

OTHER OUTCOMES:
Arterial Stiffness - Augmentation Index (AI) | Baseline and 12 weeks
  Differences in fenofibrate induced-changes in AI across rs6008845 genotypes
Haematopoietic stem/progenitor cells (HSPCs) | Baseline and 12 weeks
  Differences in fenofibrate induced-changes in circulating levels of HSPC across rs6008845 genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Luca Morieri, MD PhD, Principal Investigator — University Hospital of Padova
Locations (1):
- University Hospital of Padova, Padua, Padua, Italy

REFERENCES:
- [Background] Morieri ML, Shah HS, Sjaarda J, Lenzini PA, Campbell H, Motsinger-Reif AA, Gao H, Lovato L, Prudente S, Pandolfi A, Pezzolesi MG, Sigal RJ, Pare G, Marcovina SM, Rotroff DM, Patorno E, Mercuri L, Trischitta V, Chew EY, Kraft P, Buse JB, Wagner MJ, Cresci S, Gerstein HC, Ginsberg HN, Mychaleckyj JC, Doria A. PPARA Polymorphism Influences the Cardiovascular Benefit of Fenofibrate in Type 2 Diabetes: Findings From ACCORD-Lipid. Diabetes. 2020 Apr;69(4):771-783. doi: 10.2337/db19-0973. Epub 2020 Jan 23. PMID 31974142
- [Background] Morieri ML, Gao H, Pigeyre M, Shah HS, Sjaarda J, Mendonca C, Hastings T, Buranasupkajorn P, Motsinger-Reif AA, Rotroff DM, Sigal RJ, Marcovina SM, Kraft P, Buse JB, Wagner MJ, Gerstein HC, Mychaleckyj JC, Pare G, Doria A. Genetic Tools for Coronary Risk Assessment in Type 2 Diabetes: A Cohort Study From the ACCORD Clinical Trial. Diabetes Care. 2018 Nov;41(11):2404-2413. doi: 10.2337/dc18-0709. Epub 2018 Sep 27. PMID 30262460
- [Background] Morieri ML, Shah H, Doria A; the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Genetic Study Group. Variants in ANGPTL4 and the Risk of Coronary Artery Disease. N Engl J Med. 2016 Dec 8;375(23):2304-2305. doi: 10.1056/NEJMc1607380. No abstract available. PMID 28112899